CLINICAL TRIAL: NCT03968770
Title: A Probiotic Intervention on Pain Hypersensitivity and Microbiota Composition in Patients With Pain-osteoarthritis: Study Protocol for a Randomized Controlled Trial
Brief Title: Probiotic for Pain Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Jorge Hugo Villafañe, PhD, Researcher, Fondazione Don Carlo Gnocchi Onlus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Microbiota-PainOA
Record Dates: First submitted 2019-05-25; First posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Osteoarthritis of Multiple Joints
Keywords: Osteoarthritis; Pain; Microbiota
MeSH Terms: conditions — Osteoarthritis; Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind (Subject, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Probiotic product plus usual medical care (NSAIDs use and the promotion of a healthy lifestyle).
  Interventions: Dietary Supplement: Experimental group; Other: Usual medical care
- Control group (Placebo Comparator): Sham probiotical plus usual medical care (NSAIDs use and the promotion of a healthy lifestyle).
  Interventions: Dietary Supplement: Control group; Other: Usual medical care

INTERVENTIONS:
Dietary Supplement: Experimental group — Probiotic (Lactobacillus casei) once daily taken by 6 weeks.
  Arms: Experimental group
Dietary Supplement: Control group — Placebo of Probiotic once daily taken by 6 weeks.
  Arms: Control group
Other: Usual medical care — NSAIDs, once daily taken and promotion of a healthy lifestyle by 6 weeks.

SUMMARY:
Many people with symptomatic Osteoarthritis (OA) report chronic joint pain, especially if those patients are older than 50 years. In Europe OA is the most common form of chronic pain condition (34%) reported and entails a high economic and social burden for society. Probiotic treatment has been shown to promote bone metabolism, reduce pain and inflammatory responses of age-related musculoskeletal disorders, including OA. Gut microbiota has been proven to be of crucial importance in maintaining human health. However, the microbiota profile changes with aging, while the loss of microbiota diversity and the alterations in the optimal composition and quantity of beneficial microbes are believed to increase the risk of many diseases. Interestingly, emerging evidence leads to the hypothesis that alterations in the gut microbiome could also be considered as possible triggering factors in the onset of musculoskeletal disorders such as OA. We hypothesize that these patients with pain-OA will demonstrate an alteration of the gut microbiota to associated with the intensity of pain.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will have hip or knee OA according on radiographic findings (Kellgren-Lawrence scale ≥3) and who require and eligible for chronic, daily therapy with an NSAIDs to control OA sign and symptoms. A physiatrist (physician) will establish the diagnosis of pain-OA.

Exclusion Criteria:

* Psychiatric or neurological disorders, celiac disease, lactose intolerance, or allergies or other ongoing illnesses (i.e., irritable bowel syndrome, diabetes, ulcerative colitis, etc.) or recent antibiotic treatment (i.e., <3 months before the beginning of the study).
* Participants with known hypersensitivity to celecoxib, ibuprofen, naproxen, aspirin or esomeprazole, etc.
* Participants require treatment with aspirin > 325 mg /day.
* Participants who smoked more than 10 cigarettes per day were excluded.
* Participants will be excluded also if they score greater than 6 points on the Beck Depression Inventory (BDI) or more than 30 points in the State Trait Anxiety Inventory (STAI), dementia and not Italian speaking due to the high level of language skills required for questionnaires and quantitative sensory testing.
* Post-traumatic OA (e.g., fractures), congenital hip deformities, surgical interventions to the hip or knee, Legg-Calvé-Perthes disease, or degenerative or non-degenerative neurological conditions in which pain perception is altered will be excluded

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Change from Visual analogue scale (VAS) at 6 weeks | Baseline, immediately post-intervention (6 weeks), and follow up (4 weeks)
Change from Pressure Pain Thresholds (PPT) at 6 weeks | Baseline, immediately post-intervention (6 weeks), and follow up (4 weeks)
  PPT will be assessed bilaterally [in the center of the anterior aspect of patella (knee) and the trochanter site (hip)]
Change from Inflammatory cytokines at 6 weeks | Baseline, immediately post-intervention (6 weeks), and follow up (4 weeks)
  Fasting serum concentrations of interleukin (IL)-6, tumor necrosis factor (TNF)-α, soluble IL-6 receptor (IL-6sR), soluble IL-1 receptor (IL-1sR), and C-reactive protein (CRP) were measured by enzyme-linked immunosorbent assays.
Change from Microbiota at 6 weeks | Baseline, immediately post-intervention (6 weeks), and follow up (4 weeks)
  Microbiota composition will be identified through fecal samples for total genomic DNA extraction. The bacteria belonging to Clostridium sensu stricto, Enterobacteriaceae, Escherichia coli, Bifidobacterium, Lactobacillus and yeast were dosed using quantitative PCR approach targeted on 16S rRNA gene

CONTACTS AND LOCATIONS:
Overall Officials: Jorge H Villafañe, PhD, Principal Investigator — Fondazione Don Carlo Gnocchi Onlus

IPD SHARING:
Plan to Share IPD: No